CLINICAL TRIAL: NCT03043365
Title: Effect of Fish Oil Enriched In Omega-11 Fatty Acid On Lipoprotein Metabolism In Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 170050; 17-H-0050
Record Dates: First submitted 2017-02-03; First posted 2017-02-06 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2019-11

CONDITIONS: Lipoprotein Metabolism; PCSK9; Proteomics
Keywords: Fish Oils; Long Chain Monounsaturated Fatty Acids (LCMUFA); Lipoproteins; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Docosahexaenoic Acids; Eicosapentaenoic Acid; Fish Oils; Fatty Acids, Unsaturated

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Control Fish Oil first, then Saury Oil (Experimental): Subjects randomized to the control fish oil arm will take the equivalent to 3g of control /day (12 gel capsules/day) for 8 plus or less 2 weeks and crossover to the LCMUFA-rich saury oil capsule arm
  Interventions: Drug: control fish oil
- Arm 2: Saury Oil first, then Control Fish Oil (Experimental): Subjects randomized to the LCMUFA-rich saury oil arm will take the equivalent to 3g of control/day (12 gel capsules/day) for 8 plus or less 2 weeks and crossover to the control fish oil capsule arm
  Interventions: Drug: LCMUFA-rich saury oil
- Washout Period (No Intervention): 8 week washout period to occur between week 8 and week 16. No study supplement taken by subject at this time.

INTERVENTIONS:
Drug: control fish oil — 4 capsules, 3 times a day after meals
  Other Names: DHA, docosahexaenoic acid (DHA), eicosapentaenoic acid (EPA), EPA (fish oils); fish oils, marine oils, N3 fatty acids, omega 3 polyunsaturated fatty acid (PUFA), polyunsaturated fatty acids,; PUFA, W3 fatty acids
  Arms: Arm 1: Control Fish Oil first, then Saury Oil
Drug: LCMUFA-rich saury oil — 4 capsules, 3 times a day after meals
  Other Names: long-chain monounsaturated fatty acids
  Arms: Arm 2: Saury Oil first, then Control Fish Oil

SUMMARY:
Background:

Fish oils are known to be beneficial to health and believed to be cardio-protective. Omega-3 fatty acid is the most known fish oil available in the market. LCMUFA (long-chain monounsaturated fatty acids) is also a fish oil but it is derived from fish that consumes a diet rich in omega-11 fatty acid. Researchers want to study omega-11 fatty acid enriched fish oil and understand its effect on cardiovascular health.

Objective:

To understand the effects of LCMUFA from fish oil on cardiovascular health.

Eligibility:

Healthy volunteers ages 18 and older with no history of cardiovascular disease

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Fasting blood and urine tests
* Optional stool sample
* Questions about their diet, exercise, and the types of medicines and dietary supplements they take
* 7-day food diary
* Cardio-Ankle Vascular Index (CAVI): Blood pressure is taken in the arms and legs. The heart is monitored.
* After the screening visit, participants will take 4 gel capsules, 3 times a day after meals, for 8-10 weeks.
* Electrocardiogram (EKG)

Participants will have 3 additional visits. All include repeats of the screening tests.

Visit 2 is 8 weeks after the screening visit. Participants will stop taking the capsules for 8 weeks after this visit.

Visit 3 is at least 16 weeks after starting the supplement. Participants will take 4 capsules, 3 times a day after meals, for 8 weeks after this visit.

Visit 4 is 8 weeks after starting the second supplement.

DETAILED DESCRIPTION:
Serum cholesterol is transported by lipoproteins, such as very low-density lipoprotein (VLDL), low-density lipoproteins (LDL) and high-density lipoproteins (HDL), which vary in their relationship to cardiovascular disease risk. LDL, for example, is proatherogenic, whereas HDL is cardio-protective. Long-chain monounsaturated fatty acids (LCMUFA), fatty acids over 18 carbons in length with a single double bond, have been shown in mice to decrease proatherogenic lipoproteins, such as LDL, and reduce atherosclerosis. This study will test the hypothesis that LCMUFA supplementation in humans will favorably alter the lipoprotein lipid profile in regard to cardiovascular disease risk. In addition, we will assess other parameters related to lipoprotein composition and function, as well as other biomarkers related to coagulation and inflammation, which have previously been shown to be affected by supplementation with omega-3 fatty acids.

This clinical research project is designed as a pilot, randomized, double-blinded, crossover study that will investigate the effect of a fish oil enriched with LCMUFA on lipoprotein metabolism. Subjects will receive control fish oil enriched in oleic acid, a monounsaturated fatty acid (C18:1), or a fish oil supplement produced from Saury fish (rich in LCMUFA) for approximately 8-10 weeks, with a wash out period of 8-10 weeks between the two arms of the study. The study consists of 4 outpatient visits when laboratory or research samples and CAVI tests will be performed. A 7-day food diary, pill count, and red cell membrane fatty acid levels will be monitored to assess compliance.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Male and female participants 18 years of age or above.
* Subject must be healthy, with no known history of cardiovascular disease.
* Pre-menopausal or women of childbearing potential must be non-lactating and using an effective form of birth control during the course of the study.
* Subject understands protocol and provides written, informed consent in addition to a willingness to comply with specified follow-up evaluations.

EXCLUSION CRITERIA:

* Pregnancy, planned pregnancy (within the study period) or women currently breastfeeding.
* Subjects with weight changes greater than 20% over the past 3 months.
* Subjects planning a significant change in diet or exercise levels.
* Subjects already consuming more than 1.5 g per day of eicosapentaenoic acid (EPA) or docosahexaenoic acid (DHA) in any form.
* Known sensitivity or allergy to fish, shellfish or omega-3 fatty acids supplements
* Subjects with known bleeding disorders (for example, Hemophilia)
* Subjects previously diagnosed with atrial fibrillation
* Subjects with clinically diagnosed hepatic disease (including but not limited to auto immune disease, hepatitis and cirrhosis)
* Subjects with chronic diarrhea, gastric bypass or lap-band procedures, ostomies, bowel motility problems, or other conditions that could affect intestinal fat absorption
* Subjects with any acute and life-threatening condition, such as prior sudden cardiac arrest, acute myocardial infarction (last three months), stroke, embolism
* Liver enzymes (aspartate aminotransferase (AST) or alanine aminotransferase (ALT)) levels above 3x upper limit of normal
* Subjects with a thyroid-stimulating hormone (TSH) greater than 1.5x upper limits of normal (ULN) or clinical evidence of hypo or hyperthyroidism
* Subjects taking supplements or medications that affect lipoproteins for at least the past 8 weeks, such as fish oil supplements, bile-acid sequestrants, plant sterol supplements, fibrates, statins or Niacin.
* Subjects with hemoglobin <10g/dL
* Subject with platelet counts <60x103/microliter
* Subjects with uncontrolled hypertension (resting blood pressure > 160 mmHg systolic and /or > 100 mm Hg diastolic)
* Subject with uncontrolled diabetes (hemoglobin A1c (HbA1c) greater than or equal to 10)
* Subjects who consume excessive alcohol (binge drinking on 5 or more days in the past month)
* Subject participating in other clinical studies and/or receiving other investigational drug products prior to randomization
* Subject taking PCSK9 inhibitors within 8 weeks prior to enrollment
* Subjects being treated with tamoxifen, estrogens, or progestins that have not been stable for >4 weeks.
* Subjects initiating new medications or patients on multiple medications may also be excluded according to investigator discretion
* Anticipated surgery during the study period
* Blood donation in the last 2 weeks or planned blood donation during the study
* Subjects requiring regular transfusions for any reason
* Subjects may also be excluded for any reason that may compromise their safety or the accuracy of research data.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Amar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-seven healthy volunteers were recruited from June 2017 through March 2018 at the National Institutes of Health (NIH) (Bethesda, MD)
Groups:
- Arm 1: Control Fish Oil Arm Then Saury Oil: Subjects randomized to the control fish oil arm will take the equivalent to 3g of control /day (12 gel capsules/day) for 8 plus or less 2 weeks and cross-over to the Long Chain Monounsaturated Fatty Acids (LCMUFA)-rich saury oil capsule arm control fish oil: 4 capsules, 3 times a day after meals
- Arm 2 - Saury Oil Arm Then Control Fish Oil: Subjects randomized to the LCMUFA-rich saury oil arm will take the equivalent to 3g of control/day (12 gel capsules/day) for 8 plus or less 2 weeks and crossover to the control fish oil capsule arm Long Chain Monounsaturated Fatty Acids (LCMUFA)-rich saury oil: 4 capsules, 3 times a day after meals
Period: Weeks 0 to Week 8
Arm/Group | Arm 1: Control Fish Oil Arm Then Saury Oil | Arm 2 - Saury Oil Arm Then Control Fish Oil
Started | 20 | 17
Completed | 17 | 14
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 2 | 0
Period: Week 8 to Week 16 - Washout Period
Arm/Group | Arm 1: Control Fish Oil Arm Then Saury Oil | Arm 2 - Saury Oil Arm Then Control Fish Oil
Started | 17 | 14
Completed | 16 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Week 16 to Week 24
Arm/Group | Arm 1: Control Fish Oil Arm Then Saury Oil | Arm 2 - Saury Oil Arm Then Control Fish Oil
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Control Fish Oil First, Then Saury Oil: Subjects randomized to the control fish oil arm will take the equivalent to 3g of control /day (12 gel capsules/day) for 8 plus or less 2 weeks and crossover to the LCMUFA-rich saury oil capsule arm control fish oil: 4 capsules, 3 times a day after meals
- Arm 2:Saury Oil First, Then Control Fish Oil: Subjects randomized to the LCMUFA-rich saury oil arm will take the equivalent to 3g of control/day (12 gel capsules/day) for 8 plus or less 2 weeks and crossover to the control fish oil capsule arm LCMUFA-rich saury oil: 4 capsules, 3 times a day after meals
- Total: Total of all reporting groups
Arm/Group | Arm 1: Control Fish Oil First, Then Saury Oil | Arm 2:Saury Oil First, Then Control Fish Oil | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 37
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (12.6) | 32.3 (12.9) | 34.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in Lipid Profile at 8 Weeks
Description: The primary outcome measures of this study will be the change from baseline to end of intervention period (8 weeks) in the lipid profile (total cholesterol (TC), triglycerides (TG), high-density lipoprotein cholesterol (HDL-C), low-density lipoprotein cholesterol (LDL-C)) for the control and research supplement groups.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Arm 1 - Control Fish Oil Arm: Subjects randomized to the control fish oil arm will take 3g of control /day (12 gel capsules/day) for 8 weeks
- Arm 2 - Saury Oil Arm: Subjects randomized to the LCMUFA-rich saury oil arm will take the equivalent to 3g of control/day (12 gel capsules/day) for 8 weeks
Arm/Group | Arm 1 - Control Fish Oil Arm | Arm 2 - Saury Oil Arm
Number analyzed (Participants) | 30 | 30
mg/dL
  TG (mg/dL) | 52 (21.1) | 56.1 (26.5)
  TC (mg/dL) | 184.3 (45.6) | 181.7 (50.9)
  HDL-C (mg/dL) | 67.9 (16.9) | 68.7 (19.7)
  LDL-C (mg/dL) | 102.7 (45.2) | 98.6 (50.6)

2. Secondary Outcome: Changes Lipoprotein Particle Number, Composition and Size (sdLDL, LDL-TG, ApoE-HDL, ApoA-I, ApoB)
Description: Secondary outcome measurements will be changes in proteomics, lipoprotein particle number, high-density lipoprotein (HDL) functional test (i.e. efflux study) composition and size. Secondary outcome will measure the following: Small dense low density lipoprotein (sdLDL); Low-Density Lipoprotein Triglycerides (LDL-TG); Apolipoprotein E-containing high-density lipoprotein (ApoE-HDL); apolipoprotein A-I (ApoA-I); Apolipoprotein B (ApoB).
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Arm 1 - Control Fish Oil Arm: Subjects randomized to the control fish oil arm will take the equivalent to 3g of control /day (12 gel capsules/day) for 8 weeks
Arm/Group | Arm 1 - Control Fish Oil Arm | Arm 2 - Saury Oil Arm
Number analyzed (Participants) | 30 | 30
mg/dL
  sdLDL (mg/dL) | 29.7 (16.4) | 29 (17.9)
  LDL-TG (mg/dL) | 14.4 (6.3) | 14.7 (5.7)
  ApoE-HDL (mg/dL) | 6.3 (1.7) | 6.5 (2.1)
  ApoA-I (mg/dL) | 158.3 (26.8) | 156.1 (30.4)
  ApoB (mg/dL) | 91.4 (31.1) | 89 (33.8)

3. Secondary Outcome: Changes Lipoprotein Particle Number, Composition and Size in Oxidized Low-density Lipoprotein (oxLDL)
Description: Secondary outcome measurements will be changes in proteomics, lipoprotein particle number, high-density lipoprotein (HDL) functional test (i.e. efflux study) composition and size.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Control Fish Oil Arm | Arm 2 - Saury Oil Arm
Number analyzed (Participants) | 30 | 30
U/L | 75.3 (24.8) | 72.9 (26.1)

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Arm 1: Control Fish Oil Arm: Subjects randomized to the control fish oil arm will take the equivalent to 3g of control /day (12 gel capsules/day) for 8 weeks
- Arm 2: Saury Oil Arm: Subjects randomized to the LCMUFA-rich saury oil arm will take the equivalent to 3g of control/day (12 gel capsules/day) for 8 weeks
- Washout Period: No intervention administer to participants.
Arm/Group | Arm 1: Control Fish Oil Arm | Arm 2: Saury Oil Arm | Washout Period
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 2/34 | 2/33 | 1/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Control Fish Oil Arm (N=34) | Arm 2: Saury Oil Arm (N=33) | Washout Period (N=31)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin biopsy of left leg (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Toe Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03043365/Prot_SAP_000.pdf